CLINICAL TRIAL: NCT02524067
Title: Modified Environment for Agitation in Patients With Traumatic Brain Injury: a Controlled Multicenter
Brief Title: Modified Environment for Agitation in Patients With TBI
Acronym: ABS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Regionshospitalet Hammel Neurocenter (Other); Rigshospitalet, Denmark (Other); Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ABS project
Record Dates: First submitted 2015-07-08; First posted 2015-08-14 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2016-09

CONDITIONS: Traumatic Brain Injury (TBI); Agitated Behaviour
MeSH Terms: conditions — Brain Injuries, Traumatic; Psychomotor Agitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention (Experimental): Intervention: Circadian lighting, systematic information, music, foreclosure of the individual patient
  Interventions: Behavioral: Multifactorial circadian concept

INTERVENTIONS:
Behavioral: Multifactorial circadian concept — Circadian light, systematic information, music, individual foreclosure

SUMMARY:
This study examines the effect of an intervention consisting of dynamic circadian light and sound therapy, as well as systematic information on sleep pattern, agitated behavior and functioning level.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate and severe Traumatic Brain Injury (TBI)
* Diagnosed with Glasgow Coma Score (GCS) lower than 13-

Exclusion Criteria:

* Patients with psychiatric diagnose and not speaking danish -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-09; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Agitation on Agitated Behaviour Scale (ABS) | One year
Functional abilities on the Early Functional Abilities Scale (EFA) | One year
Functional abilities on the Glasgow Outcome Extend Scale | 12 month after admission

SECONDARY OUTCOMES:
Orientation and duration of post-traumatic amnesia on the Galveston Orientation and Amnesia Scale (GOAT) | One year

CONTACTS AND LOCATIONS:
Overall Officials: Jens Christian H Sorensen, Professor, Study Chair — Aarhus University Hoapital
Locations (1):
- Leanne Langhorn, Aarhus, Region Midt, Denmark